CLINICAL TRIAL: NCT05461209
Title: A Phase 3 Study Comparing Talquetamab to Belantamab Mafodotin in Participants With Relapsed/Refractory Multiple Myeloma Who Have Received at Least 4 Prior Therapies Including an Immunomodulatory Drug, a Proteasome Inhibitor, and an Anti-CD38 Antibody
Brief Title: A Study of Comparing Talquetamab to Belantamab Mafodotin in Participants With Relapsed/Refractory Multiple Myeloma
Acronym: MonumenTAL-5
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109235; 64407564MMY3008 (Other: Janssen Research & Development, LLC); 2022-001442-38 (EudraCT Number)
Expanded Access: NCT05503550 (No longer available)
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/ Refractory Multiple Myeloma
MeSH Terms: interventions — talquetamab; belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Talquetamab (Experimental): Participants will receive talquetamab subcutaneously (SC).
  Interventions: Drug: Talquetamab
- Arm B: Belantamab Mafodotin (Active Comparator): Participants will receive belantamab intravenously (IV).
  Interventions: Drug: Belantamab Mafodotin

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered as subcutaneous injection.
  Other Names: JNJ-64407564
  Arms: Arm A: Talquetamab
Drug: Belantamab Mafodotin — Belantamab Mafodotin will be administered as intravenous infusion.
  Arms: Arm B: Belantamab Mafodotin

SUMMARY:
The purpose of this study is to compare the efficacy of talquetamab versus belantamab mafodotin in terms of overall response rate (ORR) or progression-free survival (PFS).

DETAILED DESCRIPTION:
Multiple myeloma is an incurable, malignant, plasma cell disorder that accounts for approximately 18 percent (%) of hematological malignancies, making it the second most common hematologic malignancy. Talquetamab (also known as JNJ-64407564) is a humanized immunoglobulin G4 (IgG4) bispecific antibody designed to target G Protein-coupled receptor family C group 5 member D (GPRC5D+) cells and cluster of differentiation 3 (CD3) receptor complex on T-cells. Belantamab mafodotin is a humanized B-cell maturation antigen (BCMA)-targeting monoclonal antibody (mAb) conjugated to a cytotoxic agent maleimidocaproyl monomethyl auristatin F (MMAF) which disrupts the microtubule network, leading to cell cycle arrest and apoptosis. This study will investigate the possible improvement of ORR or PFS with talquetamab compared with belantamab mafodotin in participants with relapsed or refractory multiple myeloma who have received at least 4 prior therapies including an anti-CD38 mAb (alone or in combination), and whose disease is refractory to at least one proteasome inhibitor (PI) and one immunomodulatory drug (IMiD). The study will consists of a screening phase, treatment phase (until confirmed progressive disease, start of subsequent antimyeloma therapy, death, intolerable toxicity, withdrawal of consent, or end of the study, whichever occurs first), and post-treatment follow-up phase (until death, withdrawal of consent, loss to follow-up, or end of the study, whichever occurs first). Safety evaluations will include a review of adverse events, physical examinations, eastern cooperative oncology group (ECOG) performance status, clinical laboratory tests, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Documented multiple myeloma as defined by the criteria: a) multiple myeloma according to international myeloma working group (IMWG) diagnostic criteria b) measurable disease at screening, as assessed by central laboratory, defined by any of the following i) serum M-protein level greater than or equal to (>=) 1.0 gram per deciliter (g/dL) ii) urine M-protein level >=200 milligram (mg)/24 hours iii) Light chain multiple myeloma without measurable M-protein in the serum or the urine: serum free light chain (sFLC) >=10 milligram per deciliter (mg/dL) (central laboratory) and abnormal serum immunoglobulin kappa lambda free light chain (FLC) ratio
* Received at least 4 prior antimyeloma therapies including an anti-cluster of differentiation 38 (CD38) monoclonal antibody (mAb) (alone or in combination) and is refractory per IMWG criteria to at least one proteasome inhibitor (PI), and one immunomodulatory drug (IMiD)
* Documented evidence of progressive disease based on investigator's determination of response by IMWG criteria on or after their last regimen
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at screening
* A female participant of childbearing potential must have a negative serum pregnancy test at screening, and must agree to further serum or urine pregnancy tests during the study and within 6 months after receiving the last dose of study treatment

Exclusion Criteria:

* Contraindications or life-threatening known allergies, hypersensitivity, or intolerance to any study drug or its excipients
* Stroke or seizure within 6 months prior to signing informed consent form (ICF)
* Prior or concurrent exposure to belantamab mafodotin
* Current corneal epithelial disease except mild punctate keratopathy
* Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain magnetic resonance imaging (MRI) and lumbar cytology are required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 1 year 3 months
  ORR is defined as percentage of participants with confirmed best overall response of partial response (PR) or better according to international myeloma working group (IMWG) criteria.
Progression-free Survival (PFS) | Up to 1 year 3 months
  PFS is defined as the duration from the date of randomization to either progressive disease or death, whichever comes first.

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) or Better Response Rate | Up to 4 years
  VGPR or better response rate is defined as percentage of participants with best overall response of VGPR or better according to IMWG criteria.
Complete Response (CR) or Better Response Rate | Up to 4 years
  CR or better response is defined as percentage of participants with best overall response of CR or better according to IMWG criteria.
Overall Survival (OS) | Up to 4 years
  OS is defined as the time from randomization to date of death due to any cause.
Time to Progression on the First Subsequent Line of Therapy or Death, Whichever Comes First (PFS2) | Up to 4 years
  PFS2 is defined as time from randomization to progression on the first subsequent line of therapy or death due to any cause, whichever comes first.
Number of Participants with Adverse Events (AEs) | Up to 4 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | Up to 4 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.
Number of Participants with Abnormalities in Clinical Laboratory Assessments | Up to 4 years
  Number of participants with abnormalities in clinical laboratory assessments (such as serum chemistry and hematology [including coagulation]) will be reported.
Serum Concentration of Talquetamab | Up to 4 years
  Serum samples will be analyzed to determine concentrations of talquetamab using a validated, specific, and sensitive electrochemiluminescent immunoassay (ECLIA) method.
Number of Participants with Anti-drug Antibodies (ADAs) to Talquetamab | Up to 4 years
  Number of participants with ADAs to talquetamab will be reported.
Titers of ADAs to Talquetamab | Up to 4 years
  Titers of ADAs to talquetamab will be reported.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) | Baseline up to 4 years
  The EORTC-QLQ-C30 Version 3 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 5 single symptom items (dyspnea, insomnia, appetite loss, constipation, and diarrhea) and a single impact item (financial difficulties). The recall period is 7 days ("past week"), and responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level.
Change from Baseline in EuroQol 5-Dimension Questionnaire 5-Level (EQ-5D-5L) | Baseline up to 4 years
  EQ-5D-5L is a generic measure of health status. For purposes of this study, the EQ-5D-5L will be used to generate utility scores for use in cost-effectiveness analyses. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change from Baseline in EuroQol 5-Dimension Questionnaire 5-Level (FACT-G) | Baseline up to 4 years
  FACT-G is a 27-item questionnaire designed to measure 4 domains of HRQoL in cancer patients: physical, social, emotional, and functional well-being. In its Physical Well-Being subscale, the FACT-G includes a question concerning side effect bother (item GP5: "I am bothered by side effects of treatment"), rated on a 5-point Likert scale from "not at all" to "very much." This single item will be included as an overall summary measure of the burden of treatment toxicities compared with each other.
Time to Sustained Worsening in EORTC-QLQ-C30 | Up to 4 years
  EORTC-QLQ-C30 Version 3 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 5 single symptom items (dyspnea, insomnia, appetite loss, constipation, and diarrhea) and a single impact item (financial difficulties). The recall period is 7 days ("past week"), and responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level.
Time to Sustained Worsening in EQ-5D-5L | Up to 4 years
  The EuroQol 5-Dimension Questionnaire 5-Level (EQ-5D-5L) is a generic measure of health status. For purposes of this study, the EQ-5D-5L will be used to generate utility scores for use in cost-effectiveness analyses. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time to Sustained Worsening in FACT-G | Up to 4 years
  FACT-G is a 27-item questionnaire designed to measure 4 domains of HRQoL in cancer patients: physical, social, emotional, and functional well-being. In its Physical Well-Being subscale, the FACT-G includes a question concerning side effect bother (item GP5: "I am bothered by side effects of treatment"), rated on a 5-point Likert scale from "not at all" to "very much." This single item will be included as an overall summary measure of the burden of treatment toxicities compared with each other.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States
- Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency